CLINICAL TRIAL: NCT01152021
Title: Comparing Safety and Efficacy of Dexmedetomidine and Propofol in Patients Requiring Sedation for MRI Scanning
Brief Title: Comparing Safety and Efficacy of Dexmedetomidine and Propofol
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Publication of a similar study. Not ethical to continue.
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Randy Prescilla, Assistant in Perioperative Anesthesia, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-05-0250
Record Dates: First submitted 2010-06-25; First posted 2010-06-29 (Estimated); Results first posted 2019-05-21 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Safety and Efficacy of Sedation Medications
Keywords: dexmedetomidine; propofol; sedation; MRI; scanning; pediatric; children; Magnetic Resonance Imaging
MeSH Terms: interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine Group (Active Comparator): Dexmedetomidine given as 2mcg/kg bolus over 10 minutes followed by 1.5mcg/kg/hr infusion for duration of scan. The bolus may be repeated up to 2 times at any time during the sedation in the event that adequate sedation conditions (minimum Ramsay Sedation Score of 4) are not achieved. In the event that dexmedetomidine is unable to achieve motionless conditions, after a total of 3 boluses, 0.5 mg/kg IV pentobarbital may be administered at q1 minute intervals up to a maximum of 2 mg/kg, per established protocol.
  Interventions: Drug: Dexmedetomidine
- Propofol Group (Active Comparator): Propofol bolus at an initial dose of 1 mg/kg over 1 minute then up to two additional 1 mg/kg boluses may be administered (total 3 mg/kg) - each over a one (1) minute interval, waiting 30 seconds after completion of each bolus to reassess sedation level. Once a minimum Ramsey Sedation Score 4 is achieved, an infusion at 125 mcg/kg/min is initiated. It may be titrated to 300 mcg/kg/min. If there is movement or awakening the patient may be rebolused with no more than 2 doses of Propofol at 1 mg/kg over 1 minute, in the same dosing manner as described above, waiting 30 seconds between doses. If adequate sedation is not achieved, 0.5 mg/kg IV pentobarbital may be administered at q1 minute intervals up to a maximum of 2 mg/kg.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Dexmedetomidine — An initial bolus of 2 mcg/kg of dexmedetomidine will be administered over 10 minutes. This bolus can be repeated up to 2 times if sedation conditions are not achieved. Once successful sedation has been achieved, a 1.5 mcg/kg/hr infusion is initiated until the MRI is complete.
  Other Names: Precedex
  Arms: Dexmedetomidine Group
Drug: Propofol — An initial bolus of 1mg/kg of propofol will be administered over 1 minute. This bolus can be repeated up to 2 times if sedation conditions are not achieved. Once successful sedation has been achieved, a propofol infusion of 125 mcg/kg/min is initiated until the MRI is complete.
  Other Names: Diprivan
  Arms: Propofol Group

SUMMARY:
This is a prospective, open label randomized study. The purpose of this study is to compare propofol with dexmedetomidine for pediatric monitored anesthesia care for MRI, specifically identifying important patient demographics and looking at important outcomes including adverse events.

DETAILED DESCRIPTION:
Patients will be randomized to either arm of the study. Throughout the sedation and recovery period, all study patients will have careful, routine documentation of hemodynamics (blood pressure, heart rate, plus oximeter, respiratory rate) as well as sedation depth. Patients will remain in recovery room until they have maintained discharge criteria for 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 3 - 11 years
* Patient is scheduled for MRI at Children's Hospital Boston.
* Patient meets criteria to receive either dexmedetomidine or propofol sedation
* Patient's guardian provides written consent

Exclusion Criteria:

* Patient does not meet established sedation criteria
* Patient has history of allergy, intolerance, or reaction to dexmedetomidine or propofol or hypersensitivity
* Patient has current, repaired, or risk for Moya-Moya disease
* Patient has had a stroke within the past six months
* Patient has uncontrolled hypertension
* Patient currently uses beta antagonist, alpha 2 agonist or calcium blocker
* Known soy, Lecithin, or egg allergy

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2011-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randy Prescilla, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Propofol Group: Propofol bolus of 1 mg/kg over 1 minute then up to two additional 1 mg/kg boluses may be given (total 3 mg/kg) - each over a one (1) minute interval, waiting 30 seconds after completion of each bolus to reassess sedation level. Once a minimum Ramsey Sedation Score 4 is achieved, an infusion at 125 mcg/kg/min is initiated. It may be titrated to 300 mcg/kg/min. If there is movement or awakening the patient may be rebolused with no more than 2 doses of Propofol at 1 mg/kg over 1 minute, in the same dosing manner as described above, waiting 30 seconds between doses. If adequate sedation is not achieved, 0.5 mg/kg IV pentobarbital may be administered at q1 minute intervals up to a maximum of 2 mg/kg.
  Propofol: An initial bolus of 1mg/kg of propofol will be given over 1 minute. This bolus can be repeated up to 2 times if sedation conditions are not achieved. Once successful sedation has been achieved, a propofol infusion of 125 mcg/kg/min is initiated until the MRI is complete.
Period: Overall Study
Arm/Group | Dexmedetomidine Group | Propofol Group
Started | 8 | 7
Completed | 2 | 1
Not Completed | 6 | 6
Not completed — Adverse Event | 4 | 4
Not completed — Study drug had expired | 1 | 0
Not completed — Physician Decision | 1 | 1
Not completed — No access to study drug in Pharmacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Propofol Group: Propofol bolus at an initial dose of 1 mg/kg over 1 minute then up to 2 additional 1 mg/kg boluses may be given (total 3 mg/kg) - each over 1 minute, wait 30 seconds after bolus completion to reassess sedation level. Once a minimum Ramsey Sedation Score 4 is achieved, an infusion at 125 mcg/kg/min is initiated. It may be titrated to 300 mcg/kg/min. If there is movement or awakening the patient may be rebolused with no more than 2 doses of Propofol at 1 mg/kg over 1 minute, in the same dosing manner as described above, waiting 30 seconds between doses. If adequate sedation is not achieved, 0.5 mg/kg IV pentobarbital may be administered at q1 minute intervals up to a maximum of 2 mg/kg.
  Propofol: An initial bolus of 1mg/kg of propofol will be administered over 1 minute. This bolus can be repeated up to 2 times if sedation conditions are not achieved. Once successful sedation has been achieved, a propofol infusion of 125 mcg/kg/min is initiated until the MRI is complete.
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine Group | Propofol Group | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 7 | 15
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events During the Sedation and Recovery Period
Description: Adverse events will be described by type, system involvement and level of severity.
Time Frame: During sedation, recovery period and overnight, up to 24 hours
Measure: Number; unit: Number of events
Groups:
- Dexmedetomidine Group: Adverse events in subjects who received dexmedetomidine given bolus and infusion for duration of scan, with or without IV pentobarbital
- Propofol Group: Adverse events in subjects who received propofol bolus and infusion with or without IV pentobarbital
Arm/Group | Dexmedetomidine Group | Propofol Group
Number analyzed (Participants) | 8 | 7
Number of events | 4 | 5

2. Secondary Outcome: Clinical Parameters (Sedation Scales, Hemodynamic Variables, Clinical Observations)
Description: Sedation scores, mean arterial blood pressures, clinical observations during sedation and recovery period
Time Frame: During sedation, recovery and overnight, up to 24 hours
Population: Enrollment was slow and during enrollment for this study, a paper from Cincinnati Children Hospital Medical Center compared use of dexmedetomidine and propofol in children undergoing MRI, which answered most of the questions that this study wanted to address. With the publication of these results, the investigator decided to discontinue this study.
Groups:
- Dexmedetomidine Group: Subjects who received dexmedetomidine
- Propofol Group: Subjects who received propofol group
Arm/Group | Dexmedetomidine Group | Propofol Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Propofol Group: Propofol bolus at an initial dose of 1 mg/kg over 1 minute then up to 2 additional 1 mg/kg boluses may be given (total 3 mg/kg) - each over 1 minute interval, wait 30 seconds after bolus completion to reassess sedation level. Once a minimum Ramsey Sedation Score 4 is achieved, an infusion at 125 mcg/kg/min is initiated. It may be titrated to 300 mcg/kg/min. If there is movement or awakening the patient may be rebolused with no more than 2 doses of Propofol at 1 mg/kg over 1 minute, in the same dosing manner as described above, waiting 30 seconds between doses. If adequate sedation is not achieved, 0.5 mg/kg IV pentobarbital may be administered at q1 minute intervals up to a maximum of 2 mg/kg.
  Propofol: An initial bolus of 1mg/kg of propofol will be administered over 1 minute. This bolus can be repeated up to 2 times if sedation conditions are not achieved. Once successful sedation has been achieved, a propofol infusion of 125 mcg/kg/min is initiated until the MRI is complete.
Arm/Group | Dexmedetomidine Group | Propofol Group
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 4/8 | 4/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexmedetomidine Group (N=8) | Propofol Group (N=7)
hypotension (Blood and lymphatic system disorders) | 4 (4) | 3 (3) — Drop in Mean Arterial Pressure (MAP) > 20% of lowest awake age-adjusted norms
low pulse oximetry level (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Drop in oxygen saturation (SaO2) <95% in MRI recovery. Face mask O2 given for 17 minutes.
cluster seizures (Nervous system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated (halted prematurely) due to publication of a similar study and it was deemed unethical to continue.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes